CLINICAL TRIAL: NCT00203996
Title: Sleep, Metabolic, and Cardiovascular Dysfunction in Polycystic Ovary Syndrome
Brief Title: Polycystic Ovary Syndrome (PCOS) and Sleep Apnea
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Did not meet target patient accrual goals
Sponsor: University of Chicago (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12861B; R01HL075079 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2013-07-16 (Estimated); Last update posted 2023-03-21 (Actual); Status verified 2023-02

CONDITIONS: Polycystic Ovary Syndrome; Obstructive Sleep Apnea
Keywords: polycystic ovary syndrome; metabolic syndrome; obstructive sleep apnea; impaired glucose tolerance; insulin resistance
MeSH Terms: conditions — Polycystic Ovary Syndrome; Sleep Apnea, Obstructive; Metabolic Syndrome; Glucose Intolerance; Insulin Resistance | interventions — Continuous Positive Airway Pressure; Estrogens; Leuprolide; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (10):
- Aim 1: Placebo (No Intervention): One of the 3 treatment arms in Aim 1: Placebo. No subjects were randomized to this arm.
- Aim 1: Pioglitazone (Experimental): One of the 3 treatment arms in Aim 1: Pioglitazone. No subjects were randomized to this arm.
  Interventions: Drug: pioglitazone
- Aim 1: Leuprolide + Estrogen/Progestin (Experimental): One of the 3 treatment arms in Aim 1: depot leuprolide plus estrogen/progestin replacement. No subjects were randomized to this arm.
  Interventions: Drug: depot leuprolide plus estrogen/progestin replacement
- Aim 2: PCOS + SDB (Experimental): One of the 2 study groups in Aim 2: Women with polycystic ovary syndrome (PCOS) and sleep disordered breathing (SDB) were treated with 8 weeks of continuous positive airway pressure (CPAP).
  Interventions: Device: continuous positive airway pressure (CPAP)
- Aim 2: Matched Controls (Experimental): One of the 2 study groups in Aim 2: Women who were of similar age to those in the PCOS+SDB group were treated with 8 weeks of continuous positive airway pressure (CPAP). The recruitment of control subjects for this protocol was hindered by the difficulty in finding subjects who met both inclusion and exclusion criteria. As a consequence, the sample size of control subjects was insufficient to allow for any meaningful conclusions to be drawn. Statistical analyses were not possible due to insufficient sample size.
  Interventions: Device: continuous positive airway pressure (CPAP)
- Aim 3: REM frag - SWS supp - Baseline (Experimental): Each subject was assessed under three experimental conditions in the following order.
  REM fragmentation: Rapid eye movement (REM) sleep will be fragmented by experimentally induced microarousals for 3 consecutive nights and non-REM sleep will be left undisturbed.
  Slow wave sleep (SWS) suppression: Slow wave activity will be suppressed without awakening the subject and REM sleep will be left undisturbed.
  Baseline: "Baseline" sleep (i.e., with no experimental intervention) assessment is recorded. This assessment may have been recorded as the first, second, or third intervention.
  Interventions: Procedure: REM frag; Procedure: SWS supp
- Aim 3: REM frag - Baseline - SWS supp (Experimental): Each subject was assessed under three experimental conditions in the following order.
  REM fragmentation: Rapid eye movement (REM) sleep will be fragmented by experimentally induced microarousals for 3 consecutive nights and non-REM sleep will be left undisturbed.
  Baseline: "Baseline" sleep (i.e., with no experimental intervention) assessment is recorded. This assessment may have been recorded as the first, second, or third intervention.
  SWS suppression: Slow wave activity will be suppressed without awakening the subject and REM sleep will be left undisturbed.
  Interventions: Procedure: REM frag; Procedure: SWS supp
- Aim 3: Baseline - REM frag - SWS supp (Experimental): Each subject was assessed under three experimental conditions in the following order.
  Baseline: "Baseline" sleep (i.e., with no experimental intervention) assessment is recorded. This assessment may have been recorded as the first, second, or third intervention.
  REM fragmentation: Rapid eye movement (REM) sleep will be fragmented by experimentally induced microarousals for 3 consecutive nights and non-REM sleep will be left undisturbed.
  SWS suppression: Slow wave activity will be suppressed without awakening the subject and REM sleep will be left undisturbed.
  Interventions: Procedure: REM frag; Procedure: SWS supp
- Aim 3: SWS supp - REM frag - Baseline (Experimental): Each subject was assessed under three experimental conditions in the following order.
  SWS suppression: Slow wave activity will be suppressed without awakening the subject and REM sleep will be left undisturbed.
  REM fragmentation: Rapid eye movement (REM) sleep will be fragmented by experimentally induced microarousals for 3 consecutive nights and non-REM sleep will be left undisturbed.
  Baseline: "Baseline" sleep (i.e., with no experimental intervention) assessment is recorded. This assessment may have been recorded as the first, second, or third intervention.
  Interventions: Procedure: REM frag; Procedure: SWS supp
- Aim 3: Baseline - SWS supp - REM frag (Experimental): Each subject was assessed under three experimental conditions in the following order.
  Baseline: "Baseline" sleep (i.e., with no experimental intervention) assessment is recorded. This assessment may have been recorded as the first, second, or third intervention.
  SWS suppression: Slow wave activity will be suppressed without awakening the subject and REM sleep will be left undisturbed.
  REM fragmentation: Rapid eye movement (REM) sleep will be fragmented by experimentally induced microarousals for 3 consecutive nights and non-REM sleep will be left undisturbed.
  Interventions: Procedure: REM frag; Procedure: SWS supp

INTERVENTIONS:
Device: continuous positive airway pressure (CPAP) — CPAP is the most effective treatment available for sleep disordered breathing. CPAP provides a constant, controllable pressure to keep your upper airway open during sleep so that you can breathe normally. The pressure acts much in the same way as a splint and holds the airway open.
  Other Names: Continuous Positive Airway Pressure
  Arms: Aim 2: Matched Controls; Aim 2: PCOS + SDB
Drug: depot leuprolide plus estrogen/progestin replacement — Depot leuprolide is a long-acting, modified version of the natural brain hormone, gonadotropin releasing hormone (GnRH). This study drug will temporarily reduce the pituitary hormones that stimulate the ovaries to make both female (estrogen) and male (testosterone) hormones. The effect of this study drug will last approximately 12 weeks. During this time, your female hormone levels will be brought to normal by the use of a patch that contains estrogen and progesterone. This patch is placed on the skin and is changed twice a week. The subject will continue to wear this patch for 4 weeks after the end of the study, until the effects of the Lupron injection wear off.
  Other Names: Lupron
  Arms: Aim 1: Leuprolide + Estrogen/Progestin
Drug: pioglitazone — Pioglitazone (Actos). Pioglitazone is an oral medication approved in the Unites States for the treatment of patients with type 2 diabetes (however it is not approved for studies in this protocol). This is one of a class of drugs known as thiazolidinediones. This class of drugs has been associated with potential beneficial changes in the metabolism (use of glucose by the body) as well as lipids (fats) in the blood.
  Other Names: Actos
  Arms: Aim 1: Pioglitazone
Procedure: REM frag — Rapid eye movement (REM) sleep will be fragmented by experimentally induced microarousals for 3 consecutive nights and non-REM sleep will be left undisturbed.
  Arms: Aim 3: Baseline - REM frag - SWS supp; Aim 3: Baseline - SWS supp - REM frag; Aim 3: REM frag - Baseline - SWS supp; Aim 3: REM frag - SWS supp - Baseline; Aim 3: SWS supp - REM frag - Baseline
Procedure: SWS supp — SWS: Slow wave activity will be suppressed without awakening the subject and REM sleep will be left undisturbed.
  Arms: Aim 3: Baseline - REM frag - SWS supp; Aim 3: Baseline - SWS supp - REM frag; Aim 3: REM frag - Baseline - SWS supp; Aim 3: REM frag - SWS supp - Baseline; Aim 3: SWS supp - REM frag - Baseline

SUMMARY:
Polycystic ovary syndrome (PCOS) affects 5-10% of women in the United States. Its onset is usually at the time of puberty with manifestations of menstrual irregularity, hirsutism, and obesity. Women with PCOS suffer at an early stage of adulthood from all of the components of the metabolic syndrome, a syndrome that typically has its peak in mid-life in other subject populations. Women with PCOS are more insulin resistant than weight-matched control women and have exceptionally high rates of early-onset impaired glucose tolerance and type 2 diabetes, as well as a substantially elevated risk for hypertension, dyslipidemia, coronary, and other vascular diseases. While recent evidence indicates that the prevalence of sleep-disordered breathing (SDB) is 30-40 fold higher in PCOS than in weight-matched control women, the possible role of SDB in causing the increased metabolic and cardiovascular risks of PCOS has not been evaluated. The overall objective of the proposed study is to analyze the direction of causality between sleep disturbances and markers of the metabolic syndrome in PCOS.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) affects 5-10% of women and may be viewed as the combination of hyperandrogenism with the classical features of the metabolic syndrome in young women. PCOS presents a unique opportunity to dissect the relationship between metabolic and cardiovascular risk and sleep disordered breathing (SDB) in a population where intrinsic effects of aging have not yet developed. Because a relationship between obstructive sleep apnea, insulin resistance and elevated testosterone levels has also been observed in men and in women without PCOS, insights gained from studies in PCOS will have broad implications.

The Specific Aims of the present application are:

Specific Aim 1: to test the hypothesis that sleep disturbances are caused by hyperandrogenemia and hyperinsulinemia that characterize PCOS. Following a detailed baseline evaluation of sleep, hormonal, metabolic and cardiovascular parameters, women with PCOS will be randomized to an 8-week treatment phase with pioglitazone or depot leuprolide plus estrogen/progestin replacement or placebo. Pioglitazone will reduce insulin levels, and consequently androgen levels, in PCOS. We will compare the effects of androgen reduction alone (depot leuprolide plus estrogen/progestin) to those of insulin plus androgen reduction achieved with pioglitazone. Primary comparisons will be the change in sleep parameters from baseline between: placebo & pioglitazone; placebo & leuprolide/estrogen/progestin; pioglitazone & leuprolide/estrogen/progestin.

Specific Aim 2: to test the hypothesis that sleep disturbances cause the hormonal, metabolic and cardiovascular alterations seen in women with PCOS. PCOS women with SDB and matched control women with SDB will be evaluated at baseline and following 8 weeks of CPAP treatment. The primary comparison will be between baseline and post-treatment parameters in PCOS women. The secondary comparison will be the post-treatment change from baseline between PCOS and control women to test the hypothesis that for the same degree in improvement in SDB, the magnitude of change in metabolic and cardiovascular measures will be greater in PCOS than in controls.

Specific Aim 3: to test the hypothesis that in normal young women, experimental manipulation of sleep that recapitulates the sleep disturbances characteristic of women with PCOS will result in metabolic, hormonal, and cardiovascular alterations that are typical of the metabolic syndrome. A group of healthy young women will be studied twice using a randomized cross-over design. In one study, rapid eye movement (REM) sleep will be fragmented by experimentally induced microarousals for 3 consecutive nights and non-REM sleep will be left undisturbed. In the other, slow wave activity will be suppressed without awakening the subject and REM sleep will be left undisturbed. Each study will be preceded by 2 nights of baseline sleep. Results were not reported for Aim 3 since no devices or drugs were tested in this aim.

ELIGIBILITY:
Inclusion Criteria:

* PCOS subjects will be recruited from the Endocrinology Clinics of the University of Chicago. All will be at least 2 years post-menarche and less than 40 years of age. A diagnosis of PCOS will require:

  * the presence of oligo/amenorrhea;
  * hyperandrogenemia, defined by a supranormal plasma free testosterone level (> 10 pg/ml);
  * hyperandrogenism, as evidenced by infertility, hirsutism, acne, or androgenetic alopecia; and
  * exclusion of nonclassic 21-hydroxylase deficiency congenital adrenal hyperplasia, Cushing's syndrome, hypothyroidism, or significant elevations in serum prolactin. Thus, all subjects will meet the National Institutes of Health (NIH) consensus criteria for PCOS.
* Control subjects will be matched, as closely as possible, for age, ethnicity, body mass index (BMI), and body fat distribution [as assessed by single cut abdominal computed tomography (CT) scan and dual energy x-ray absorptiometry (DEXA) scan].
* Normal lean (BMI <25 kg/m2) women will be between 18 and 40 years of age, in good health, with normal menstrual cycles, no sleep complaints, no history of endocrine disorder. All studies will be initiated in the early follicular phase (days 2-4).

Exclusion Criteria:

* For at least 2 months before the study, all subjects (PCOS and control) must not take steroid preparations (including oral contraceptives), medications known to alter insulin secretion and/or action, or medications known to influence sleep.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2003-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Ehrmann, M.D., Principal Investigator — University of Chicago; Esra Tasali, M.D., Study Director — University of Chicago; Eve Van Cauter, Ph.D., Study Director — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Result] Tasali E, Chapotot F, Leproult R, Whitmore H, Ehrmann DA. Treatment of obstructive sleep apnea improves cardiometabolic function in young obese women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2011 Feb;96(2):365-74. doi: 10.1210/jc.2010-1187. Epub 2010 Dec 1. PMID 21123449
- [Result] Tasali E, Leproult R, Ehrmann DA, Van Cauter E. Slow-wave sleep and the risk of type 2 diabetes in humans. Proc Natl Acad Sci U S A. 2008 Jan 22;105(3):1044-9. doi: 10.1073/pnas.0706446105. Epub 2008 Jan 2. PMID 18172212
- [Derived] Tasali E, Van Cauter E, Hoffman L, Ehrmann DA. Impact of obstructive sleep apnea on insulin resistance and glucose tolerance in women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2008 Oct;93(10):3878-84. doi: 10.1210/jc.2008-0925. Epub 2008 Jul 22. PMID 18647805

RESULTS

PARTICIPANT FLOW:
Groups:
- Aim 1: Leuprolide + Estrogen/Progestin: One of the 3 treatment arms in Aim 1: Leuprolide + estrogen/progestin replacement. No subjects were randomized to this arm.
- Aim 2: PCOS + SDB With CPAP: One of the 2 study groups in Aim 2: Women with polycystic ovary syndrome (PCOS) and sleep disordered breathing (SDB) were treated with 8 weeks of continuous positive airway pressure (CPAP).
- Aim 2: Matched Controls With CPAP: One of the 2 study groups in Aim 2: Women who were of similar age to those in the PCOS+SDB group were treated with 8 weeks of continuous positive airway pressure (CPAP).
- Aim 3: REM Frag - SWS Supp - Baseline: Each subject was assessed under three experimental conditions in the following order.
  REM fragmentation: Rapid eye movement (REM) sleep will be fragmented by experimentally induced microarousals for 3 consecutive nights and non-REM sleep will be left undisturbed.
  SWS suppression: Slow wave activity will be suppressed without awakening the subject and REM sleep will be left undisturbed.
  Baseline: "Baseline" sleep (i.e., with no experimental intervention) assessment is recorded. This assessment may have been recorded as the first, second, or third intervention.
Period: Overall Study
Arm/Group | Aim 1: Placebo | Aim 1: Pioglitazone | Aim 1: Leuprolide + Estrogen/Progestin | Aim 2: PCOS + SDB With CPAP | Aim 2: Matched Controls With CPAP | Aim 3: REM Frag - SWS Supp - Baseline | Aim 3: REM Frag - Baseline - SWS Supp | Aim 3: Baseline - REM Frag - SWS Supp | Aim 3: SWS Supp - REM Frag - Baseline | Aim 3: Baseline - SWS Supp - REM Frag
Started | 0 | 0 | 0 | 19 | 4 | 3 | 2 | 4 | 2 | 3
Aim 3 Only: First Intervention | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 4 | 2 | 3
Aim 3 Only: Washout | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 2 | 2
Aim 3 Only: Second Intervention | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 2 | 2
Aim 3 Only: Second Washout | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 2 | 2
Aim 3 Only: Third Intervention | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 2 | 2
Completed | 0 | 0 | 0 | 9 | 3 | 3 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 10 | 1 | 0 | 0 | 2 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 6 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — CPAP machine malfunction | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Scheduling issue | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Aim 3: All Participants: Includes groups randomized to any experimental ordering in Aim 3
- Total: Total of all reporting groups
Arm/Group | Aim 1: Placebo | Aim 1: Pioglitazone | Aim 1: Leuprolide + Estrogen/Progestin | Aim 2: PCOS + SDB With CPAP | Aim 2: Matched Controls With CPAP | Aim 3: All Participants | Total
Number analyzed (Participants) | 0 | 0 | 0 | 19 | 4 | 14 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] |  |  |  | 31.2 (5.3) | 32.2 (5.8) | 24.6 (2.7) | 28.8 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  |  |  | 19 | 4 | 5 | 28
  Male |  |  |  | 0 | 0 | 9 | 9

OUTCOME MEASURES:

1. Primary Outcome: Aim 1: Apnea-Hypopnea Index (AHI) [Baseline]
Description: Apnea-hypopnea index (AHI) is an index used to assess the severity of sleep apnea based on the total number of complete cessations (apnea) and partial obstructions (hypopnea) of breathing occurring per hour of sleep.
Time Frame: baseline
Population: No participants were randomized to these study arms.
Arm/Group | Aim 1: Placebo | Aim 1: Pioglitazone | Aim 1: Leuprolide + Estrogen/Progestin
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Aim 1: Apnea-hypopnea Index (AHI) [After Treatment]
Description: as for outcome 1
Time Frame: 8 weeks
Population: No participants were randomized to these study arms.
Arm/Group | Aim 1: Placebo | Aim 1: Pioglitazone | Aim 1: Leuprolide + Estrogen/Progestin
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Aim 2: Insulin Sensitivity Index (SI) From Intravenous Glucose Tolerance Test [Baseline]
Description: Insulin sensitivity Index (SI) is the increase in net fractional glucose clearance rate per unit change in plasma insulin concentration after an intravenous glucose load. SI quantifies the capacity of insulin to promote glucose disposal.
Time Frame: baseline (0 weeks)
Population: The recruitment of control subjects for this protocol was hindered by the difficulty in finding subjects who met both inclusion and exclusion criteria. As a consequence, the sample size of control subjects was insufficient to allow for any meaningful conclusions to be drawn. Statistical analyses were not possible due to insufficient sample size.
Measure: Mean (Standard Error); unit: mU/(liter x min)
Arm/Group | Aim 2: PCOS + SDB With CPAP | Aim 2: Matched Controls With CPAP
Number analyzed (Participants) | 9 | 3
mU/(liter x min) | 0.87 (0.13) | 3.67 (1.01)

4. Primary Outcome: Aim 2: Insulin Sensitivity Index (SI) From Intravenous Glucose Tolerance Test [After CPAP]
Description: as for outcome 3
Time Frame: 8 weeks
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mU/(liter x min)
Arm/Group | Aim 2: PCOS + SDB With CPAP | Aim 2: Matched Controls With CPAP
Number analyzed (Participants) | 9 | 3
mU/(liter x min) | 0.93 (0.17) | 2.57 (0.34)

5. Secondary Outcome: Aim 1: Blood Pressure [Baseline]
Description: Blood pressure is the pressure of blood within the arteries, produced primarily by the contraction of the heart muscle.
Time Frame: baseline (0 weeks)
Population: No participants were randomized to these study arms.
Arm/Group | Aim 1: Placebo | Aim 1: Pioglitazone | Aim 1: Leuprolide + Estrogen/Progestin
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Aim 1: Blood Pressure [After Treatment]
Description: Blood pressure is the pressure of blood within the arteries, produced primarily by the contraction of the heart muscle.
Time Frame: 8 weeks
Population: No participants were randomized to these study arms.
Arm/Group | Aim 1: Placebo | Aim 1: Pioglitazone | Aim 1: Leuprolide + Estrogen/Progestin
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Aim 1: Visceral Adiposity [Baseline]
Description: Visceral adiposity refers to the degree of fat located in the peritoneal cavity (abdominal area) that surrounds the body's internal organs.
Time Frame: up to half of an hour
Population: No participants were randomized to this arm.
Arm/Group | Aim 1: Placebo | Aim 1: Pioglitazone | Aim 1: Leuprolide + Estrogen/Progestin
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Aim 1: Visceral Adiposity [After Treatment]
Description: as for outcome 7
Time Frame: up to half of an hour
Population: No participants were randomized to this arm.
Arm/Group | Aim 1: Placebo | Aim 1: Pioglitazone | Aim 1: Leuprolide + Estrogen/Progestin
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Aim 2: Mean Cortisol Levels Over 24 Hours, Per Patient [Baseline]
Description: This outcome is defined as the average concentration of cortisol (a glucocorticoid produced by the adrenal gland) in the blood, measured repeatedly over a 24 hour period in each patient individually.
Time Frame: 10 minutes, over a period of 24 hours
Population: as for outcome 3
Measure: Mean (Standard Error); unit: microgram/deciliter
Arm/Group | Aim 2: PCOS + SDB With CPAP | Aim 2: Matched Controls With CPAP
Number analyzed (Participants) | 9 | 3
microgram/deciliter | 8.6 (0.9) | 6.1 (0.2)

10. Primary Outcome: Aim 2: Acute Insulin Resistance to Intravenous Glucose (AIRg) [Baseline]
Description: Acute insulin resistance to intravenous glucose (AIRg) is a measure of the secretion of insulin during the first 10 minutes after an intravenous glucose load. AIRg addresses adequacy of insulin secretion.
Time Frame: baseline (0 weeks)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mU/(liter x min)
Arm/Group | Aim 2: PCOS + SDB With CPAP | Aim 2: Matched Controls With CPAP
Number analyzed (Participants) | 9 | 3
mU/(liter x min) | 1711 (370) | 695 (228)

11. Primary Outcome: Aim 2: Acute Insulin Resistance to Intravenous Glucose (AIRg) [After CPAP]
Description: as for outcome 10
Time Frame: 8 weeks
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mU/(liter x min)
Arm/Group | Aim 2: PCOS + SDB With CPAP | Aim 2: Matched Controls With CPAP
Number analyzed (Participants) | 9 | 3
mU/(liter x min) | 1614 (385) | 722 (211)

12. Secondary Outcome: Aim 2: Mean Cortisol Levels Over 24 Hours, Per Patient [After Treatment]
Description: as for outcome 9
Time Frame: 10 minutes, over a period of 24 hours
Population: as for outcome 3
Measure: Mean (Standard Error); unit: microgram/deciliter
Arm/Group | Aim 2: PCOS + SDB With CPAP | Aim 2: Matched Controls With CPAP
Number analyzed (Participants) | 9 | 3
microgram/deciliter | 7.8 (0.5) | 6.5 (0.2)

13. Secondary Outcome: Aim 2: Mean Leptin Levels Over 24 Hours, Per Patient [Baseline]
Description: This outcome is defined as the average concentration of leptin (a hormone produced by the fat cells that affects feeding behavior and appetite) in the blood, measured repeatedly over a 24 hour period in each patient individually.
Time Frame: 15 minutes over a period of 24 hours
Population: as for outcome 3
Measure: Mean (Standard Error); unit: nanogram/milliliter
Arm/Group | Aim 2: PCOS + SDB With CPAP | Aim 2: Matched Controls With CPAP
Number analyzed (Participants) | 9 | 3
nanogram/milliliter | 67.6 (10.5) | 56.9 (1.6)

14. Secondary Outcome: Aim 2: Mean Leptin Levels Over 24 Hours, Per Patient [After Treatment]
Description: as for outcome 13
Time Frame: 15 minutes over a period of 24 hours
Population: as for outcome 3
Measure: Mean (Standard Error); unit: nanogram/milliliter
Arm/Group | Aim 2: PCOS + SDB With CPAP | Aim 2: Matched Controls With CPAP
Number analyzed (Participants) | 9 | 3
nanogram/milliliter | 65.8 (9.9) | 57.4 (2.3)

15. Primary Outcome: Aim 3: Insulin Sensitivity Index (SI) From Intravenous Glucose Tolerance Test [Baseline]
Description: as for outcome 3
Time Frame: Baseline
Population: Due to technical issues, REM fragmentation data were not analyzable. Technical issues also resulted in non-analyzable data for two subjects in the SWS suppression study, thereby decreasing the sample size from 11 to 9 subjects.
Measure: Mean (Standard Error); unit: mU/(liter x min)
Groups:
- Aim 3: REM Fragmentation: Rapid eye movement (REM) sleep will be fragmented by experimentally induced microarousals for 3 consecutive nights and non-REM sleep will be left undisturbed.
- Aim 3: SWS Suppression: Slow wave sleep (SWS) suppression: Slow wave activity will be suppressed without awakening the subject and REM sleep will be left undisturbed.
Arm/Group | Aim 3: REM Fragmentation | Aim 3: SWS Suppression
Number analyzed (Participants) | 0 | 9
mU/(liter x min) |  | 8.42 (1.12)

16. Primary Outcome: Aim 3: Insulin Sensitivity Index (SI) From Intravenous Glucose Tolerance Test [After 3 Nights of SWS Suppression]
Description: as for outcome 3
Time Frame: 3 nights
Population: as for outcome 15
Measure: Mean (Standard Error); unit: mU/(liter x min)
Arm/Group | Aim 3: REM Fragmentation | Aim 3: SWS Suppression
Number analyzed (Participants) | 0 | 9
mU/(liter x min) |  | 5.87 (0.74)

ADVERSE EVENTS:
Groups:
- Aim 3: SWS Suppression: SWS: Slow wave activity will be suppressed without awakening the subject and REM sleep will be left undisturbed.
Arm/Group | Aim 1: Placebo | Aim 1: Pioglitazone | Aim 1: Leuprolide + Estrogen/Progestin | Aim 2: PCOS + SDB With CPAP | Aim 2: Matched Controls With CPAP | Aim 3: REM Fragmentation | Aim 3: SWS Suppression
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/19 | 0/4 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 1/19 | 0/4 | 0/14 | 0/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aim 1: Placebo (N=0) | Aim 1: Pioglitazone (N=0) | Aim 1: Leuprolide + Estrogen/Progestin (N=0) | Aim 2: PCOS + SDB With CPAP (N=19) | Aim 2: Matched Controls With CPAP (N=4) | Aim 3: REM Fragmentation (N=14) | Aim 3: SWS Suppression (N=14)
Vaginal bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 — Abnormal vaginal bleeding is any vaginal bleeding unrelated to normal menstruation.

LIMITATIONS AND CAVEATS:
No participants were randomized to any of the 3 study arms in Aim 1. Also, the recruitment of control subjects for Aim 2 was hindered by the difficulty in finding subjects who met both inclusion and exclusion criteria.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes